CLINICAL TRIAL: NCT00002653
Title: VIIITH MYELOMATOSIS TRIAL: A RANDOMISED TRIAL OF TREATMENT FOR INDUCING FIRST PLATEAU PHASE ABCM VS 3 COURSES OF ABCM FOLLOWED BY ORAL WEEKLY CYCLOPHOSPHAMIDE
Brief Title: Combination Chemotherapy With or Without Cyclophosphamide and Prednisone in Treating Older Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064187; MRC-LEUK-MYEL-VIII; EU-94031
Record Dates: First submitted 1999-11-01; First posted 2003-04-10 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2002-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Carmustine; Cyclophosphamide; Doxorubicin; Melphalan; Prednisone; Radiotherapy

INTERVENTIONS:
Drug: carmustine
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: melphalan
Drug: prednisone
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is most effective in treating older patients with multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without cyclophosphamide and prednisone in treating older patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of doxorubicin, carmustine, cyclophosphamide, and melphalan (ABCM) with or without oral cyclophosphamide and prednisone as induction for the first plateau phase in elderly patients with previously untreated multiple myeloma.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center.

Patients receive doxorubicin IV followed immediately by carmustine IV over 1-2 hours on day 1 and oral melphalan (L-PAM) and oral cyclophosphamide (CTX) on days 22-25 (ABCM). Treatment continues every 6 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients whose blood counts recover within 6 weeks after beginning L-PAM and CTX during course 3 are randomized to 1 of 2 treatment arms. Patients whose blood counts fail to recover within 6 weeks after beginning L-PAM and CTX during course 3 are assigned to arm II.

* Arm I: Patients continue ABCM for a maximum of 12 courses in the absence of a plateau phase after completion of at least 4 courses, disease progression, or unacceptable toxicity.
* Arm II: Patients receive oral cyclophosphamide once weekly and oral prednisone every other day. Treatment continues every 6 weeks in the absence of a plateau phase after completion of 3 courses of ABCM plus a minimum of 8 weeks on arm II or less than 3 courses of ABCM plus 6 months on arm II, disease progression, or unacceptable toxicity.

Patients on both arms with bone pain or failure to respond to chemotherapy may undergo minimal radiotherapy. Patients achieving plateau phase may enter the MRC trial of interferon alfa-2b.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued for this study within approximately 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma, defined by at least 2 of the following conditions:

  * Neoplastic cell infiltrate and/or microplasmacytomas by bone marrow sections or smears

    * Plasma cell infiltrates greater than 20% of marrow nucleated cells or, if less than 20%, objective evidence of monoclonality of the plasma cells required
  * Paraprotein in blood or urine
  * Definite lytic bone lesions (not osteoporosis)
* Nonsecretory disease allowed in the presence of 1 of the following conditions:

  * Microplasmacytomas
  * Monoclonal plasmacytosis with immunoglobulin light-chain expression in cytoplasm
* No equivocal myelomatosis, defined by the following criteria:

  * Minimal or no symptoms attributable to myelomatosis
  * Pretransfusion hemoglobin greater than 10 g/dL
  * Post-hydration creatinine less than 1.47 mg/dL
  * No osteolytic lesions except minimal lesions that do not threaten pathological fracture and are not associated with pain
  * Plasma cells less than 30% of marrow nucleated cells and marrow showing normal hematopoietic activity
  * Serum beta-2 microglobulin less than 4 mg/L
  * Less than 1 g of free light-chain excretion per 1 g of creatinine
  * No objective factors indicating progressive myelomatosis

PATIENT CHARACTERISTICS:

Age:

* 65 to 74
* If under 65, higher priority is given to protocol MRC-LEUK-MYEL-VII unless entry into this study would be more appropriate

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Neutrophil count at least 1,300/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Not specified

Renal:

* See Disease Characteristics

Other:

* Ability to tolerate fluid intake of at least 3 L/day beginning at least 2 days before study entry
* Afebrile and free of infection
* No contraindication to therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior or concurrent prednisolone at 30 mg/m2/day or less (or equivalent doses of other corticosteroids) for relief of fluid-unresponsive hypercalcemia allowed

Radiotherapy:

* Prior or concurrent minimal local radiotherapy to relieve persistent bone pain or cord compression allowed

Surgery:

* Not specified

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1993-09

CONTACTS AND LOCATIONS:
Overall Officials: M. T. Drayson, MD, Study Chair — MRC Myelomatosis Trials Office
Locations (1):
- MRC Myelomatosis Trials Office, Birmingham, England, United Kingdom